CLINICAL TRIAL: NCT03023176
Title: Protective Mechanisms Against a Pandemic Respiratory Virus: B-cell, T-cell, and General Immune Response to Seasonal Influenza Vaccine. Year 5, 2013
Brief Title: T-cell And General Immune Response to Seasonal Influenza Vaccine (SLVP018) Year 5, 2013
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SU-17219-2013; 2U19AI057229-06 (NIH)
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: Trivalent, inactivated influenza vaccine; Child identical twins; Child fraternal twins
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy 1-8 year-old twins (Other): Healthy 1-8 yr old identical and fraternal twin pairs given trivalent, inactivated influenza (Fluzone® standard IIV3 0.5ml or Fluzone® standard IIV3 Pediatric Dose) per participant age and standard of care.
  Interventions: Biological: Fluzone® standard IIV3; Biological: Fluzone® standard IIV3 Pediatric Dose

INTERVENTIONS:
Biological: Fluzone® standard IIV3 — Influenza Virus Vaccine Suspension (0.5ml) for Intramuscular Injection
Biological: Fluzone® standard IIV3 Pediatric Dose — Influenza Virus Vaccine Suspension (0.25ml) for Intramuscular Injection

SUMMARY:
This study will investigate markers, mechanisms and define general predictors for immunological health by comparing influenza vaccine responses in monozygotic and dizygotic twins.

DETAILED DESCRIPTION:
The investigators plan to study the immune response to different influenza vaccines much more broadly and deeply across different age groups and with different vaccine modalities and to probe the influence of genetics on these responses using monozygotic and dizygotic twins. The investigators plan to compare various immunological responses, identify age-specific biomarkers or clusters of markers, quantify the frequency of influenza-specific T-cells pre- and post-vaccination, and determine the effective breadth of T-cell repertoire to an influenza vaccine within an individual as a function of age and to what degree this is genetically determined.

The study will be conducted in healthy young identical and fraternal 1-8 year-old twins. All participants will be immunized with seasonal trivalent inactivated influenza vaccine (IIV3). Blood samples to conduct the assays described will be taken at pre-immunization, Days 6-8 and 28 post-immunization for children requiring 1 dose of vaccine. For children requiring 2 doses of vaccine, a second immunization will be given at least 28 days after Dose 1 with responses measured on Day 6-8 and Day 28-32 post-second immunization.

Children 35 months and under will receive Fluzone® standard IIV3 Pediatric Dose, while children 36 months and older will receive Fluzone® standard IIV3.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy, twin children age 1-8 years (identical or fraternal twin pairs)
2. Parent willing to sign the informed consent form and child willing to sign assent if indicated.
3. Availability for follow-up for the planned duration of the study at least 28 days after last immunization.
4. Acceptable relevant medical history and vital signs.

Exclusion Criteria:

1. Prior off-study vaccination with trivalent inactivated influenza vaccine (IIV3) or live attenuated influenza vaccine (LAIV) in Fall 2013
2. Allergy to egg or egg products, or to vaccine components or thimerosal (if IIV3 multidose vials used)
3. Life-threatening reactions to previous influenza vaccinations
4. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
5. History of immunodeficiency (including HIV infection)
6. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
7. Chronic Hepatitis B or C
8. Recent or current use of immunosuppressive medication, including glucocorticoids (corticosteroid nasal sprays, topical steroids are permissible). History of any cancer.
9. Autoimmune disease including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
10. History of blood dyscrasias, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
11. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin.
12. Receipt of blood or blood products within the past 6 months or planned receipt of blood products prior to completion of study visits.
13. Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
14. Receipt of inactivated vaccine 14 days prior to enrollment, or planned non-study vaccination prior to completion of Visit 03 or 04 (~Day 28 after the last study vaccination)
15. Receipt of a live, attenuated vaccine within 30 days prior to first vaccination, or planned immunization with a live, attenuated vaccine before completion of study visits (inform study staff of any non-study vaccinations received during the study period).
16. Need for allergy immunization (that cannot be postponed) during the study period.
17. History of Guillain-Barre Syndrome
18. Use of investigational agents within 30 days prior to enrollment or planned use of investigational agents prior to completion of study visits.
19. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Dekker, MD, Principal Investigator — Stanford University; Mark Davis, PhD, Principal Investigator — Stanford University; Garry Nolan, PhD, Principal Investigator — Stanford University; Ann Arvin, MD, Principal Investigator — Stanford University; Stephen Quake, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Gars M, Kay AW, Bayless NL, Aziz N, Dekker CL, Swan GE, Davis MM, Blish CA. Increased Proinflammatory Responses of Monocytes and Plasmacytoid Dendritic Cells to Influenza A Virus Infection During Pregnancy. J Infect Dis. 2016 Dec 1;214(11):1666-1671. doi: 10.1093/infdis/jiw448. Epub 2016 Sep 21. PMID 27655870

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy 1-8 Year-old Twins
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy 1-8 Year-old Twins
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.06 (1.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Influenza Vaccine
Time Frame: Day 0 to 32
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy 1-8 Year-old Twins
Number analyzed (Participants) | 20
Participants | 20

2. Secondary Outcome: Number of Participants With Related Adverse Events
Time Frame: Day 0 to 32 post-immunization
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy 1-8 Year-old Twins
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Time Frame: Day 0 to 32
Description: Clinical Assessment performed at each visit
Arm/Group | Healthy 1-8 Year-old Twins
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No